CLINICAL TRIAL: NCT04528095
Title: Sequential Multiple-Assignment Randomized Trials to Compare Antipsychotic Treatments in Treatment-Resistant Schizophrenia
Brief Title: SMART Design to Compare Antipsychotic Treatments in Treatment-Resistant Schizophrenia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: TRS-SMART
Record Dates: First submitted 2020-08-12; First posted 2020-08-27 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Treatment-resistant Schizophrenia
Keywords: Schizophrenia; Treatment-resistant; Antipsychotics; Combination
MeSH Terms: conditions — Schizophrenia, Treatment-Resistant; Schizophrenia | interventions — Clozapine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Clozapine (Experimental): Clozapine 400 ~ 600mg/d or plasma concentration >350ng/ml
  Interventions: Drug: Clozapine
- Clozapine+Amisulpride (Experimental): Clozapine 400 ~ 600mg/d or plasma concentration >350ng/ml Amisulpride 200-800mg/d
  Interventions: Drug: Clozapine
- Clozapine+Gingke biloba (Experimental): Clozapine 400 ~ 600mg/d or plasma concentration >350ng/ml Gingke biloba 120-360mg/d
  Interventions: Drug: Clozapine
- MECT (Experimental): MECT:The treatment lasted for 4 months,16 times in total
  Interventions: Device: MECT
- MST (Experimental): MST:The treatment lasted for 4 months,16 times in total
  Interventions: Device: MECT
- DBS (Experimental): Two electrode emplacement groups (target nucleus accumbens and hippocampus respectively)
  Interventions: Device: DBS

INTERVENTIONS:
Drug: Clozapine — Clozapine 400 ~ 600mg/d or plasma concentration >350ng/ml Amisulpride 200-800mg/d Gingke biloba 120-360mg/d
  Other Names: Clozapine+Amisulpride; Clozapine+Gingke biloba
  Arms: Clozapine; Clozapine+Amisulpride; Clozapine+Gingke biloba
Device: MECT — MECT:The treatment lasted for 4 months,16 times in total MST:The treatment lasted for 4 months,16 times in total
  Other Names: MST
  Arms: MECT; MST
Device: DBS — Two electrode emplacement groups (target nucleus accumbens and hippocampus respectively)
  Arms: DBS

SUMMARY:
The project intends to take treatment-resistant schizophrenia as the research object and uses sequential multiple assignment randomized trial(SMART) design to define the treatment recommendations of different drug regimen for treatment resistant schizophrenia and to determine the physical enhancement regimen for clozapine-resistant schizophrenia and to explore targeted regulation scheme for ultra-resistant schizophrenia.

DETAILED DESCRIPTION:
This trial is a sequential multiple-assignment RCT design of antipsychotic drugs, planning to recruit 162 people with treatment-resistant schizophrenia followed for 12 months. The study includes three treatment phases and a naturalistic follow-up phase. Participants who meet the response criteria remain on that treatment for the duration of 12-month treatment. If the participants fail the treatment or can't tolerant the side effects, the patient moves to the next phase of the study to receive a new treatment.

ELIGIBILITY:
Inclusion Criteria:

1. meet the DSM-5 diagnostic criteria for schizophrenia,
2. be 18-55 years of age,
3. treatment-resistant schizophrenia:no response to sufficient doses (400-600 mg/ day CPZ equivalent) of at least two antipsychotics in the past 5 years,
4. Informed consent.

Exclusion Criteria:

1. Patients with medical or psychiatric comorbidities and those who require concomitant other medications are excluded.
2. Patients with contraindications to even one of the proposed treatment arms are excluded.
3. Patients with risks such as extreme agitation, stupor or suicide are excluded.
4. Female patients with pregnancy or breast-feeding are also excluded.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 162 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Response rate | Change from baseline PANSS score at 12 weeks
  25% or greater change in Positive and Negative Syndrome Scale (PANSS)

SECONDARY OUTCOMES:
Adverse reactions | baseline, 4 weeks, 8 weeks, 12 weeks, 14 weeks, 16 weeks,32 weeks
  The Barnes Akathisia Scale (BAS) (0,14,higher scores mean a worse outcome),
Adverse reactions | baseline, 4 weeks, 8 weeks, 12 weeks, 14 weeks, 16 weeks,32 weeks
  Simpson-Angus Extrapyramidal Side Effects Scale (SAS) (0,40,higher scores mean a worse outcome)
Adverse reactions | baseline, 4 weeks, 8 weeks, 12 weeks, 14 weeks, 16 weeks,32 weeks
  Abnormal Involuntary Movement Scale (AIMS) (0,42,higher scores mean a worse outcome)
Neurocognitive assessments and social function | baseline, 6 weeks, 3 months, 6 months, 9 months, 12 months
  The University of California, San Diego (UCSD) Performance- based Skills Assessment-Brief (UPSA-B) (0,100,higher scores mean a better outcome) is used to evaluate the social function,
Neurocognitive assessments and social function | baseline, 6 weeks, 3 months, 6 months, 9 months, 12 months
  The MATRICS consensus cognitive battery (MCCB) has been widely used to evaluate cognitive deficits in schizophrenia patients(0%,100%,higher scores mean a better outcome)
Clinical assessements | baseline, 4 weeks, 8 weeks, 12 weeks, 14 weeks, 16 weeks,32 weeks
  PANSS (30,210,higher scores mean a worse outcome),
Clinical assessements | baseline, 4 weeks, 8 weeks, 12 weeks, 14 weeks, 16 weeks,32 weeks
  Clinician-Rated Dimensions of Psychosis Symptom Severity (CRDPS) (0,32,higher scores mean a worse outcome),
Clinical assessements | baseline, 4 weeks, 8 weeks, 12 weeks, 14 weeks, 16 weeks,32 weeks
  Calgary Depression Scale for Schizophrenia (CDSS) (0,27,higher scores mean a worse outcome)
Clinical assessements | baseline, 4 weeks, 8 weeks, 12 weeks, 14 weeks, 16 weeks,32 weeks
  Clinical Global Impression Scale-Severity (CGI-S) (0,7,higher scores mean a worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Dengtang Liu, MD, Study Chair — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China